CLINICAL TRIAL: NCT04963959
Title: A Study on the Collection of Peripheral Blood Mononuclear Cells From Healthy Volunteers for UCAR T Production and Clinical Investigation
Brief Title: PBMC Collection for Production of UCAR T Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CT0590-CG6011
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Blood Mononuclear Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy donor (Other)
  Interventions: Device: Peripheral blood mononuclear cell apheresis

INTERVENTIONS:
Device: Peripheral blood mononuclear cell apheresis — mononuclear cell donation for tumor immunotherapy study of UCAR-T cells

SUMMARY:
The objective of the study is to collect peripheral blood mononuclear cells (PBMC) from healthy volunteers for the research and production of UCAR T cells used for Clinical trails.

DETAILED DESCRIPTION:
The study is a single-center study.

1. Screening period: All volunteers are required to sign a written informed consent form for the study; after the signing of informed consent form, the demographic data and medical history of the volunteers will be collected, and physical examinations and local laboratory tests will be performed to assess the eligibility of the volunteers. Volunteers who meet all the inclusion criteria and do not meet any exclusion criteria will receive peripheral venous whole blood sampling, and the volunteers receiving apheresis based on the assessment results will be enrolled.
2. Apheresis period: 25 volunteers who meet the inclusion criteria will undergo collection of peripheral blood mononuclear cells (PBMC) by means of apheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who signed informed consent form
2. Age ≥ 18 years and ≤ 40 years, male or female, Han nationality.
3. Weight: male ≥ 50 kg, female ≥ 45 kg; 18.5 ≤ BMI ≤ 30.
4. Temperature: 36.3-37.2℃ (Forehead temperature).

Exclusion Criteria:

1. Those with known respiratory, circulatory, digestive, urinary, blood, immune, endocrine disorders or metabolic disorders, neurological diseases, mental illnesses and those with a family history;
2. Those with known chronic skin diseases, especially infectious, allergic or inflammatory systemic skin diseases;
3. Those with known allergic diseases or recurrent allergies;
4. Those with known malignant tumors or health-affecting benign tumors;
5. Two or more physical examination results of blood pressure have shown (except for white coat hypertension): systolic blood pressure < 90 or ≥140mmHg, or diastolic blood pressure < 60 or ≥ 90 mmHg, or pulse pressure < 30 mmHg, heart rate: < 60 beats/min or >100 beats/min;
6. Laboratory tests: hemoglobin is abnormal and has clinical significant; liver and kidney function are higher than the normal upper limit and have clinical significance; 12-lead ECG is abnormal and has clinical significance, or abdominal ultrasound is abnormal and has clinical significance, or chest X-ray is abnormal and has clinical significance; abnormal coagulation function; increased CRP;
7. Those with active or latent hepatitis B or active hepatitis C, or Treponema pallidum antibody, or human immunodeficiency virus antibody, or anti-EBV IgM antibody, or anti-CMV IgM antibody, or COVID-19 DNA ;
8. Recipients of allogeneic tissue and organ or hematopoietic stem cell transplants;
9. Those who have undergone resection of vital internal organs such as stomach, kidney, spleen and lung;
10. Those who have undergone minor surgery within last 3 months, such as appendectomy and ophthalmic surgery; those who have undergone major surgery within 1 year, such as surgical treatment for gynecological benign tumors or superficial benign tumors;
11. Women who are pregnant, or have an abortion within last 6 months or gave childbirth within 1 year;
12. Those whose upper respiratory tract infection has recovered for less than 1 week, or pneumonia has recovered for less than 3 months;
13. Those whose acute pyelonephritis has recovered for less than 3 months, or those with acute exacerbation of urinary calculi;
14. Those who have been injured or wound-contaminated by equipment contaminated by blood or tissue fluids, or who have got a tattoo for less than 1 year;
15. Those who have received whole blood and blood component transfusion within 1 year;
16. Those who have received the last dose of live attenuated vaccines within 2 weeks, or have received the last dose of rubella live vaccine within 4 weeks;
17. Those who have received the last dose of rabies vaccines after being bitten by an animal within 1 year;
18. Those who have received the last dose of antitoxin or immune serum injection within 4 weeks, or those who have received the last dose of hepatitis B human immunoglobulin injection within 1 year;
19. Those who have participated in clinical trials within 3 months, or try to participate in other intervention trials during the study.
20. Those who are considered by the investigator as unsuitable for participating in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The number of peripheral blood mononuclear cells (PBMC | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No